CLINICAL TRIAL: NCT05748249
Title: "Randomized, Controlled 3-arm Clinical Study to Evaluate the Efficacy of Supplementation With Vertistop® D and Vertistop® L in Preventing Recurrences of Highly Recurring BPPV (Benign Paroxysmal Positional Vertigo)".
Brief Title: Evaluation of the Efficacy of Vertistop® D and Vertistop® L in the Prevention of BPPV Recurrence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Picciotti Pasqualina Maria, Principal Investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: VERT-2017-001
Record Dates: First submitted 2023-02-10; First posted 2023-02-28 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Benign Paroxysmal Positional Vertigo; Vitamin D; Antioxidants
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- First arm Vertistop® L. (Active Comparator): BPPV patients will be assigned to the first arm have a "sufficient" serum concentration of Vitamin D between 31 and 100 ng/mL (76 and 250 nmol/L), which will be treated with Vertistop® L.
  Interventions: Drug: Vertistop® D
- Second arm No Therapy (No Intervention): BPPV patients will be assigned to the second arm having serum concentrations of Vitamin D "Sufficient" between 31 and 100 ng/mL that will not be treated
- Third arm Vertistop® D (Experimental): In the third arm, patients with serum values of Vitamin D "insufficient" i.e. between 20 and 30 ng/mL (50- 75 nmol/L) or "deficient" i.e. less than 20 ng/mL (50 nmol/L) which they will instead be treated with Vertistop® D.
  Interventions: Drug: Vertistop® D

INTERVENTIONS:
Drug: Vertistop® D — Vitamin D supplementation
  Other Names: Vertistop® L
  Arms: First arm Vertistop® L.; Third arm Vertistop® D

SUMMARY:
The study involves the evaluation of 3 groups of subjects (3-arm study). Patients diagnosed with BPPV and "sufficient" serum concentrations of Vitamin D (>30 ng/mL, >75 nmol/L) at baseline may be treated with 2 tablets per day (morning and evening) of Vertistop® L ( Alpha-lipoic acid, carnosine, zinc and curcumin) or untreated, on the basis of the randomization criterion to which they will be assigned. Patients with Vitamin D "deficiency" (<20 ng/mL, <50 nmol/L) or Vitamin D "insufficient" (20-30 ng/mL, 50-75 nmol/L) at baseline, or subsequent follow-up, they will be treated for 2 months with Vertistop® D (alpha-lipoic acid, carnosine and zinc, vitamin D3 and vitamins of the B complex) taking 1 tablet a day (before meals).

The main purpose of the study is to evaluate, over a period of 6 months, the efficacy of Vertistop® D and Vertistop® L supplementation in preventing recurrences of BPPV (Benign Paroxysmal Positional Vertigo), in relation to blood levels of Vitamin D.

DETAILED DESCRIPTION:
Patients will be assigned to one of the three study groups following a randomization list with reference to groups 1 and 2 and according to the serum concentrations of 25(OH) Vitamin D, evaluated at the baseline visit, with reference to group 3.

The determination of the Vitamin D concentration will be requested by the Investigating physician and the report will be evaluated during the randomisation visit (V1), Visit 2, (after 2 months from enrollment/start of treatment), Visit 3 (Follow-up visit up to 4 months from enrollment) and finally Visit 4 (Follow-up visit 6 months after enrollment).

The blood sample and the Vitamin D dosage will be carried out the week before the day of the visit agreed with the Investigator, in a trusted laboratory of the patient, provided that it has the legal authorizations and the analytical methodology satisfactory the measurement intervals reported in Protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of both sexes, aged between 18 and 85 years, diagnosed with primary BPPV.
2. Patients who have BPPV of the posterior semicircular canal (SPC) geo and apo, lateral semicircular canal (SLC) geo and apo (single-canal, multi-canal).
3. Patients with relapsing BPPV, defined as two or more episodes in the past six months, or three or more episodes in the last 12 months.
4. Patients able to understand and follow the requirements of the Study Protocol and to provide their informed consent.

Exclusion Criteria:

1. Patients under the age of 18.
2. Secondary BPPV. Other causes of possible high recurrence BPPV and/or massive otolithic detachment:

   * Migraine;
   * Meniere's or delayed endolymphatic hydrops;
   * Lindsay Hemenway syndrome;
   * Otological and/or dental implant surgery in the last 3 months;
   * Conclusion within 30 days.
3. Patients with Vitamin D values exceeding 100 ng/mL (>250 nmol/L).
4. Pregnant or lactating women, as reported by the patient.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the number of BPPV recurrences in patients treated with Vertistop® D | 6 months
  Clinical Vestibular evaluation (presence of positional Nystagmus)

SECONDARY OUTCOMES:
Increased normalization of Vitamin D | 6 months
  Vitamin D evaluation

OTHER OUTCOMES:
Evaluation of BPPV recurrences in patients treated with Vertistop® L. | 6 months
  Clinical vestibular evaluation (presence of positional Nystagmus)

CONTACTS AND LOCATIONS:
Overall Officials: Pasqualina M Picciotti, Principal Investigator — Università Cattolica del Sacro Cuore, Fondazione Policlinico Gemelli IRCCS
Locations (1):
- Clinica Otorinolaringoiatrica, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bhattacharyya N, Gubbels SP, Schwartz SR, Edlow JA, El-Kashlan H, Fife T, Holmberg JM, Mahoney K, Hollingsworth DB, Roberts R, Seidman MD, Steiner RW, Do BT, Voelker CC, Waguespack RW, Corrigan MD. Clinical Practice Guideline: Benign Paroxysmal Positional Vertigo (Update). Otolaryngol Head Neck Surg. 2017 Mar;156(3_suppl):S1-S47. doi: 10.1177/0194599816689667. PMID 28248609
- [Result] Imai T, Takeda N, Ikezono T, Shigeno K, Asai M, Watanabe Y, Suzuki M; Committee for Standards in Diagnosis of Japan Society for Equilibrium Research. Classification, diagnostic criteria and management of benign paroxysmal positional vertigo. Auris Nasus Larynx. 2017 Feb;44(1):1-6. doi: 10.1016/j.anl.2016.03.013. Epub 2016 May 9. PMID 27174206
- [Result] Epley JM. Positional vertigo related to semicircular canalithiasis. Otolaryngol Head Neck Surg. 1995 Jan;112(1):154-61. doi: 10.1016/S0194-59989570315-2. PMID 7816450
- [Result] von Brevern M, Radtke A, Lezius F, Feldmann M, Ziese T, Lempert T, Neuhauser H. Epidemiology of benign paroxysmal positional vertigo: a population based study. J Neurol Neurosurg Psychiatry. 2007 Jul;78(7):710-5. doi: 10.1136/jnnp.2006.100420. Epub 2006 Nov 29. PMID 17135456
- [Result] Eggers SDZ, Bisdorff A, von Brevern M, Zee DS, Kim JS, Perez-Fernandez N, Welgampola MS, Della Santina CC, Newman-Toker DE. Classification of vestibular signs and examination techniques: Nystagmus and nystagmus-like movements. J Vestib Res. 2019;29(2-3):57-87. doi: 10.3233/VES-190658. PMID 31256095
- [Result] Buki B, Ecker M, Junger H, Lundberg YW. Vitamin D deficiency and benign paroxysmal positioning vertigo. Med Hypotheses. 2013 Feb;80(2):201-4. doi: 10.1016/j.mehy.2012.11.029. Epub 2012 Dec 14. PMID 23245911
- [Result] Sheikhzadeh M, Lotfi Y, Mousavi A, Heidari B, Bakhshi E. The effect of serum vitamin D normalization in preventing recurrences of benign paroxysmal positional vertigo: A case-control study. Caspian J Intern Med. 2016 Summer;7(3):173-177. PMID 27757201
- [Result] Taneja MK, Taneja V. Vitamin d deficiency in e.N.T. Patients. Indian J Otolaryngol Head Neck Surg. 2013 Jan;65(1):57-60. doi: 10.1007/s12070-012-0603-9. Epub 2012 Dec 1. PMID 24381922
- [Result] Elmoursy MM, Abbas AS. The role of low levels of vitamin D as a co-factor in the relapse of benign paroxysmal positional vertigo (BPPV). Am J Otolaryngol. 2021 Nov-Dec;42(6):103134. doi: 10.1016/j.amjoto.2021.103134. Epub 2021 Jun 19. PMID 34166965